CLINICAL TRIAL: NCT00148707
Title: Phase II Study of CT-2103 in Patients With Metastatic Breast Cancer
Brief Title: Study of Xyotax (CT-2103) in Patients With Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other); Brigham and Women's Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04-299
Record Dates: First submitted 2005-09-07; First posted 2005-09-08 (Estimated); Last update posted 2007-12-21 (Estimated); Status verified 2007-12

CONDITIONS: Breast Cancer; Metastatic Breast Cancer
Keywords: Metastatic Breast Cancer; HER2-negative Breast Cancer; CT-2103; Xyotax
MeSH Terms: conditions — Breast Neoplasms | interventions — paclitaxel poliglumex

INTERVENTIONS:
Drug: CT-2103 (Xyotax)

SUMMARY:
The purpose of this study is to collect information on what effects (good or bad) CT-2103 (Xyotax) has on breast cancer as well as any side effects the drug may cause.

DETAILED DESCRIPTION:
* Patients will be given CT-2103 intravenously every 3 weeks. One week after the first dose of CT-2103 a physical exam, blood work and assessment of any side effects will be performed.
* Prior to each injection of CT-2103, a physical exam, blood work and assessment of any side effects will be performed (every 3 weeks).
* Every 6 weeks the patient's cancer will be re-evaluated with either a CT scan or MRI to determine whether the treatment is working.
* Additional blood work will be performed once per week after the first two doses of CT-2103.
* The participation in this study will last at least 2 cycles (6 weeks), however patients may remain on the study as long as there is no disease progression, and they are able to tolerate the study drug without severe side effects.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of invasive breast cancer, Stage IV disease
* Age greater than 18 years
* At least one measurable target lesion as defined by RECIST that has not been previously treated with local therapy
* HER2-negative breast cancer
* Up to one prior chemotherapy for advanced or metastatic disease
* ECOG performance status 0-1
* Life expectancy > 12 weeks
* Adequate liver and bone marrow function: AST < 2.5 x ULN; Bilirubin < 1.5 x ULN; ANC > 1,500/ul; platelet count > 100,000/ul; normal PT and PTT
* At least 2 weeks since prior radiation and recovered from treatment-related toxicity

Exclusion Criteria:

* Prior taxanes for treatment of metastatic disease
* Pregnant of breast-feeding women
* HER2-positive breast cancer
* More than 1 prior chemotherapy regimen for metastatic disease
* Untreated brain metastases
* Concurrent radiotherapy or investigational drug
* Prior bone marrow or stem cell transplant
* History of other malignancy within the last 5 years, not including curatively-treated carcinoma in situ of the cervix or non-melanoma skin cancer
* Uncontrolled infection
* Active bleeding, or history of bleeding requiring transfusion
* Active cardiac disease
* Serious medical or psychiatric illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45
Dates: Start 2004-10; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
To evaluate the response to CT02103 as first or second-line treatment in patients with metastatic breast cancer.

SECONDARY OUTCOMES:
To evaluate the side effects of CT-2103 in patients with metastatic breast cancer
to evaluate the proportion of patients that have complete or partial response or stable disease at 4 months
to determine the time to progression and overall survival of patients treated with CT2103.

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence N. Shulman, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts